CLINICAL TRIAL: NCT04784403
Title: SCREENING AND SEROEPIDEMIOLOGY OF SARS-CoV-2 INFECTION AT THE UNIVERSITY OF BARCELONA: A CROSS-SECTIONAL STUDY
Acronym: UB-GTMS-COVID
Status: Completed | Type: Observational
Sponsor: Dr. Francisco Ciruela Alférez (Other)
Collaborators: Gerencia Territorial del Área Metropolitana Sur - Instituto Catalán de la Salud (Unknown); Hospital Universitario de Bellvitge (Unknown); Fundació IDIBELL (Unknown)
Responsible Party: Sponsor-Investigator, Dr. Francisco Ciruela Alférez, Sponsor's representative, University of Barcelona
Organization: University of Barcelona (Other)
Other Study IDs: UB-EPI-2020-01
Record Dates: First submitted 2020-12-21; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: SARS-CoV-2 Infection
Keywords: SARS-COV-2; prevalence; Associated factors; University of Barcelona
MeSH Terms: conditions — COVID-19 | interventions — Serologic Tests

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Students and workers at the University of Barcelona: The study population will be randomly selected from the different groups of the University:
  * Students from the different centers and type of studies (undergraduate / graduate).
  * Administrative and service personnel.
  * Teaching and Research Staff.
  Interventions: Diagnostic Test: SARS-CoV-2 PCR and serology tests

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 PCR and serology tests — Once the informed consent has been signed, the selected subjects must complete an epidemiological survey and go to a UB sample collection center to perform a PCR and serology test for SARS-CoV-2.
  Other Names: epidemiological survey

SUMMARY:
BACKGROUND: On January 7, 2020, the Chinese authorities identified as the agent responsible for the cases of atypical pneumonia of unknown etiology a new type of virus of the Coronaviridae family that has subsequently been named SARS-CoV-2, whose genetic sequence was shared by Chinese authorities on January 12 (taxonomy ID: 2697049). On January 30, 2020, the director general of the World Health Organization (WHO), following the advice of the Emergency Committee convened in accordance with the International Health Regulations (2005), declared that the COVID-19 outbreak started in Wuhan, China in December 2019, being a public health emergency of international concern. On March 11, the WHO declared the global SARS-CoV-2 pandemic.

So far, in the absence of effective vaccines or antiviral drugs, efforts have focused on identifying cases and their contacts. Both the cases and their contacts are isolated for about 14 days with the intention of minimizing the spread of this infection and avoiding an increase in the number of affected.

At the time of writing this new version of the protocol, we are immersed in the second wave of the COVID-19 pandemic. The projections of the natural history of the disease and the estimates of possible infections by SARS-CoV-2, carried out at the end of the first wave, made it possible to determine the feasibility of this second wave with the onset of cold from the autumn.

Given this scenario, the University of Barcelona, together with the Gerencia Territorial del Área Metropolitana Sud, has planned to carry out, a study of seroprevalence and screnning of SARS-CoV-2 in the population of Universidad de Barcelona users.

The results of this study will help to make preventive decisions in the face of SARS-CoV-2 infection at the UB, in relation to its teaching and administrative activities. In addition, this cross-sectional study can serve as the base study for a future follow-up study.

HYPOTHESIS: The incidence of SARS-CoV-2 infection in the group of students and workers at the University of Barcelona is similar to the incidence in the general population.

MAIN OBJECTIVE:

* Estimate the incidence of SARS-CoV-2 infection in the UB community.
* Estimate the SARS-CoV-2 seroprevalence infection in the UB community.

DETAILED DESCRIPTION:
BACKGROUND: On January 7, 2020, the Chinese authorities identified as the agent responsible for the cases of atypical pneumonia of unknown etiology a new type of virus of the Coronaviridae family that has subsequently been named SARS-CoV-2, whose genetic sequence was shared by Chinese authorities on January 12 (taxonomy ID: 2697049).

On January 30, 2020, the director general of the World Health Organization (WHO), following the advice of the Emergency Committee convened in accordance with the International Health Regulations (2005), declared that the COVID-19 outbreak started in Wuhan, China in December 2019, being a public health emergency of international concern. On March 11, the WHO declared the global SARS-CoV-2 pandemic.

So far, in the absence of effective vaccines or antiviral drugs, efforts have focused on identifying cases and their contacts. Both the cases and their contacts are isolated for about 14 days with the intention of minimizing the spread of this infection and avoiding an increase in the number of affected.

At the level of microbiological clinical practice, the diagnosis of SARS-CoV-2 infection can be made by:

1. Detection of the presence of the target nucleic acid sequences in the RNA of SARS-CoV-2 (RdRP gene of SARSCoV-2 and gene N and Orf1ab present in SARS and SARSCoV-2, gene E of SARS) in the Patient specimen by reverse transcriptase polymerase chain reaction (RT-PCR).
2. Detection of antibodies: total immunoglobulins and IgG.

At the time of writing this new version of the protocol, the country is immersed in the second wave of the COVID-19 pandemic. The projections of the natural history of the disease and the estimates of possible infections by SARS-CoV-2, carried out at the end of the first wave, made it possible to determine the feasibility of this second wave with the onset of cold from the autumn. Some of the factors that supported this hypothesis are:

1. At the end of the first wave, herd immunity against the virus was not reached. The results of the ENE-COVID study, published in the Lancet magazine in July this year, indicated that in our environment only 6% have achieved immunity.
2. Many respiratory viruses have a seasonal behavior and their circulation increases in the autumn and winter months. This is why a similar behavior was assumed in this new SARS-CoV-2 virus, experiencing greater transmissibility with the drop in temperature and increase in humidity, typical of winter periods.
3. Observing the evolution of the 1918 pandemic flu, the first wave was in 1918, but this was followed by a second and third wave, in 1919 and 1920 respectively. However, the second wave presented the peculiarity of being triggered in other areas where the first wave had not been so intense.

Given this scenario, the University of Barcelona, together with the Gerencia Territorial del Área Metropolitana Sud, has planned to carry out, a study of seroprevalence and screnning of SARS-CoV-2 in the population of UB users. The results of this study will help to make preventive decisions in the face of SARS-CoV-2 infection at the UB, in relation to its teaching and administrative activities. In addition, this cross-sectional study can serve as the base study for a future follow-up study.

HYPOTHESIS: The incidence of SARS-CoV-2 infection in the group of students and workers at the University of Barcelona is similar to the incidence in the general population.

The seroprevalence of SARS-CoV-2 infection in the group of students and workers at the University of Barcelona is similar to the seroprevalence of the general population.

MAIN OBJECTIVE

* Estimate the incidence of SARS-CoV-2 infection in the UB community.
* Estimate the SARS-CoV-2 seroprevalence infection in the UB community.

SECONDARY OBJECTIVES

Clinical objectives:

* Estimate the factors associated with the incidence in the UB community.
* Estimate the factors associated with seroprevalence in the UB community

STUDY DESIGN Cross-sectional study with epidemiological information to determine the incidence and prevalence of SARS-CoV-2 infection in the UB population, by PCR and serology tests to detect antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Adult population (18 years or more), of both sexes.
* Person linked (with identification card) to the University of Barcelona.
* Acceptance to participate in the study.

Exclusion Criteria:

There are no exclusion criteria.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The target population of this study is made up of students and workers at the University of Barcelona:
  * Students from the different centers and type of studies (undergraduate / graduate).
  * Administrative and service personnel.
  * Teaching and Research Staff.
Sampling Method: Probability Sample
Enrollment: 3356 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
Number of people with a positive SARS-CoV-2 PCR. | one day
Incidence of people with a positive SARS-CoV-2 PCR. | one day
Number of people with a positive total immunoglobulin titer and positive IgG for SARS-CoV-2. | one day
Prevalence of people with a positive total immunoglobulin titer and positive IgG for SARS-CoV-2. | one day

SECONDARY OUTCOMES:
Number of people with a positive SARS-CoV-2 Ig total titer and a negative IgG. | one day

OTHER OUTCOMES:
Estimation of associated factors ith the main variable (age, sex, university group and variables of exposure and preventive measures) | one day

CONTACTS AND LOCATIONS:
Overall Officials: Sebastià Videla Cés, MD PhD, Study Director — Hospital Universitario de Bellvitge; Esteve Fernández Muñoz, Professor, Study Director — Universidad de Barcelona
Locations (1):
- Francisco Ciruela Alférez, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pollan M, Perez-Gomez B, Pastor-Barriuso R, Oteo J, Hernan MA, Perez-Olmeda M, Sanmartin JL, Fernandez-Garcia A, Cruz I, Fernandez de Larrea N, Molina M, Rodriguez-Cabrera F, Martin M, Merino-Amador P, Leon Paniagua J, Munoz-Montalvo JF, Blanco F, Yotti R; ENE-COVID Study Group. Prevalence of SARS-CoV-2 in Spain (ENE-COVID): a nationwide, population-based seroepidemiological study. Lancet. 2020 Aug 22;396(10250):535-544. doi: 10.1016/S0140-6736(20)31483-5. Epub 2020 Jul 6. PMID 32645347
- [Background] 5. Albert Bosch. SARS-CoV-2: ¿No solo un virus? Ciclo de webinars. Patógenos Online. Grupo Especializado en Biología de Microrganismos Patógenos (GEBMP). Sociedad Española de Microbiología, 30 de junio de 2020.
- See also: Scientific-technical information report on coronavirus disease, COVID-19 in Spain. Center for Coordination of Health Alerts and Emergencies. July 3, 2020. — https://www.mscbs.gob.es/profesionales/saludPublica/ccayes/alertasActual/nCov-China/documentos/ITCoronavirus.pdf
- See also: Situation report Nro. 168 about coronavirus disease (COVID-19). World Health Organization. 16 July 2020. — https://www.who.int/docs/default-source/coronaviruse/situation-reports/20200817-weekly-epi-update-1.pdf?sfvrsn=b6d49a76_4